CLINICAL TRIAL: NCT05433766
Title: Exploring the Feasibility of the OKKO Health App to Monitor and Predict the Decline in Vision Caused by Age-related Macular Degeneration
Brief Title: Patient-centred Smartphone AI for Protecting Vision in Macular Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: OKKO Health (Industry)
Collaborators: INNOVATEUK (Unknown); Nottingham University Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); The Macular Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: OKHR-06
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2022-12

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Macular disease is the leading cause of blindness in the UK and age-related macular degeneration must undergo monitoring to determine if an injection into the eye is required that month [required in 50% of visits] - these patients are the 'frequent fliers' within ophthalmology units, visiting specialist hospital clinics on a monthly or bi-monthly basis. This project aims to create a home-monitoring algorithm that could in the future, enable the movement of 'monitoring' of chronic eye disease into the patients' homes: remotely identifying who does need an in-person appointment, and who can safely stay away from hospital.

DETAILED DESCRIPTION:
The OKKO Health application is a CE-marked medical software application that aims to monitor visual function, track symptoms and treatment, and improve patient knowledge about their condition.

To monitor visual function, OKKO implements quick and engaging activities to assess visual function, contrast sensitivity, and hyperacuity. The aim of this is to develop the app to see if it is possible to detect changes in visual function in a timely manner. This would enable regular monitoring for disease progression and/or the response of visual function to treatments between clinical visits. Home monitoring may reveal information that may support the early diagnosis of worsening conditions and may enable a greater understanding of disease progression or stabilisation. Currently unpublished data collected using the OKKO Health app highlights its acceptability when collecting visual acuity compared to gold standard techniques used in clinical practice.

OKKO includes self-monitoring features which may result in an increased (disease) awareness including vision changes between clinic visits. OKKO offers symptom and treatment tracking functionality as well as education modules to increase literacy about the disease and treatment. These elements may improve the patient's self-efficacy, enable patient empowerment, and may increase the involvement of patients in their care and more thorough communication with ophthalmologists including shared decision-making processes. Thus, these psychological and behavioural changes may alleviate the patient's burden.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with wet (neovascular) AMD in at least on eye at the start of their anti-VGEF treatment.
* Participants with wet AMD in at least one eye undergoing anti-VGEF therapy.
* Access to a device running a compatible software

  * Apple device running iOS 12 or later,
  * Android devices running Android 7.0 or later,
* Ability to read and understand English.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Vision worse than 6/60 or 1.0 LogMAR in both eyes.
* Significant cognitive impairment.
* Patients who do not have the manual dexterity to tap a screen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with macular degeneration undergoing anti-VEGF treatment, at either Queens Medical Centre, Nottingham University Hospitals NHS Trust or Oxford Eye Hospital at Oxford University Hospitals NHS Trust will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in visual status | 12 months continuous use
  Generate an algorithm to detect a change in visual status (in particular a deterioration) in advance of in-person hospital appointment.

SECONDARY OUTCOMES:
Impact of the OKKO Health app on Health literacy | 3-6 months of app use
  The HLS-EU-Q16, a validated questionnaire, will be used to assess Health Literacy at baseline and following 3-6 months of app use.
Patient engagement with OKKO Health app | 12 months continuous use
  Patient engagement will be determined through an analyses of engagement collected within the OKKO Health. Volunteers will be asked to use the OKKO Health app three times per week.
To explore the correlation of varying demographic and lifestyle factors on AMD disease progression | 12 months continuous use
  This will include identifying the correlation between the trend in the OKKO Health app data versus lifestyle data (this will include physical activity (steps taken, distance walked) and sleep recorded through the participants device). Correlations between health data (BMI and blood pressure) and OKKO Health trend data will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Foss, D.M, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford